CLINICAL TRIAL: NCT06380348
Title: A Randomized, Open-label, Parallel-controlled Phase 3 Study of Combination JMT101 and Osimertinib Compared With Cisplatin -Pemetrexed in Patients With EGFR Exon 20ins Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: JMT101 in Combination With Osimertinib, Versus Cisplatin-pemetrexed in Participants With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Characterized by Epithermal Growth Factor Receptor (EGFR) Exon 20ins Mutations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-012
Record Dates: First submitted 2024-04-09; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Local Advanced or Metastatic NSCLC
Keywords: Harboring EGFR 20ins mutation; Without prior systemic therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMT101 combined with Osimertinib (Experimental)
  Interventions: Drug: JMT101 Injection; Drug: Osimertinib tablet
- Cisplatin combined with pemetrexed (Active Comparator): Participants randomized into chemotherapy arm can receive up to 4 cycles of pemetrexed + cisplatin (pemetrexed 500 mg/m^2 + cisplatin 75mg/m^2, IV infusion, every 3 weeks) as the initial treatment. Participants whose disease has not progressed after 4 cycles of first-line platinum-based doublet chemotherapy may receive pemetrexed maintenance monotherapy until a treatment discontinuation criterion is met.
  Interventions: Drug: Cisplatin injection; Drug: Pemetrexed injection

INTERVENTIONS:
Drug: JMT101 Injection — JMT101 Injection, 6 mg/kg intravenously, over 90 mins every 14 days
  Arms: JMT101 combined with Osimertinib
Drug: Osimertinib tablet — Osimertinib 160mg once po everyday
  Arms: JMT101 combined with Osimertinib
Drug: Cisplatin injection — Cisplatin 75mg/m^2, IV infusion, on day-1 at every cycle of 21days, 4 cycles at most.
  Arms: Cisplatin combined with pemetrexed
Drug: Pemetrexed injection — Pemetrexed 500mg/m^2, IV infusion, on day-1 at every cycle of 21 days.
  Arms: Cisplatin combined with pemetrexed

SUMMARY:
This is a multicenter, randomized, open-label, parallel-controlled phase 3 study. This study aims to evaluate the efficacy and safety of JMT101 combined with Osimertinib compared with Cisplatin combined with pemetrexed in participants with local advanced or metastatic non-small-cell lung cancer harboured EGFR 20ins mutation without prior systemic therapy.

Primary objective of this study is to assess the efficacy of JMT101 combined with Osimertinib versus Cisplatin combined with pemetrexed using by （Independent Review Center）IRC-assessed Progression Free Survival (PFS) per RECIST 1.1 as primary endpoint. Approximately 398 participants are estimated to be randomized into the study. Participants enrolled will be randomized to JMT101 or Cisplatin chemotherapy in a 1:1 manner, stratified by baseline brain metastasis (with/without) and Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) (0 versus 1).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old.
2. Histologically or cytologically confirmed diagnosis of NSCLC, locally advanced (Stage IIIB and IIIC according to the 8th edition of the IASLC TNM staging criteria) or metastatic (Stage IV), not suitable for curative therapy. For central laboratory confirmation of EGFR exon 20 insertion mutation with tumour tissue/blood sample.
3. At least 1 measurable lesion per RECIST Version 1.1
4. Life expectancy ≥ 12 weeks
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
6. Adequate organ and hematologic function

Exclusion Criteria:

1. Prior treatment with any systemic anti-cancer therapy for locally advanced or metastatic NSCLC.
2. Central nervous system metastasis with associated symptom and signs.
3. Concurrent EGFR mutations: exon 19 deletion, L858R, T790M, G719X, S768I, or L861Q.
4. History of interstitial lung disease, or infectious pneumonitis need heavy antibiotics therapy
5. As judged by the investigator, unsuitable for attending the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2027-03-26 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as assessed by Independent Review Center (IRC) per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 35 months after the first participant is randomized
Overall Response Rate (ORR) by IRC per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized
Duration of Response (DoR) by IRC per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized
PFS by investigator per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized
ORR by investigator per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized
DoR by investigator per RECIST 1.1 | Up to approximately 35 months after the first participant is randomized

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Cancer Prevention and Treatment Center of Sun Yat sen University

IPD SHARING:
Plan to Share IPD: No